CLINICAL TRIAL: NCT00887783
Title: Induction Chemotherapy With Carboplatin and Navelbine Oral(R) Followed by Concomitant Navelbine Oral(R) and Irradiation in Local-regionally Advanced Non-small Cell Lung Cancer. A Randomized Phase II Study.
Brief Title: Navelbine And Radiotherapy in Locally Advanced Lung Cancer
Acronym: NARLAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); Vejle Hospital (Other); Rigshospitalet, Denmark (Other); Aalborg University Hospital (Other); Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Olfred Hansen, MD, Professor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.01
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Induction chemotherapy; Non-small cell lung cancer; Randomized phase II study; Navelbine Oral (R); 3D-conformal radiotherapy; Chemo-radiotherapy; Local-regionally advanced non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine

STUDY DESIGN:
Masking Description: No blinding after randomization
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B: 66Gy/33F+Navelbine oral 150 mg q3w (Experimental): Navelbine oral 150 mg of Vinorelbine administered in 3 weekly doses a week for 6-6½ weeks concomitant with curatively intended irradiation to 66 Gy (2 Gy x 30, 5 F á weeks).
  Radiation technique: 3D, 4D og VMAT techniques. The patients all had 2 cycles of carboplatin and vinorelbine before randomization
  Interventions: Drug: Navelbine; Radiation: 66 Gy/33F
- A: 60Gy/30F+Navelbine oral 150 mg q3w (Active Comparator): Navelbine oral 150 mg of Vinorelbine administered in 3 weekly doses a week for 6-6½ weeks concomitant with curatively intended irradiation to 60 Gy (2 Gy x 30, 5 F á weeks) Radiation technique: 3D, 4D og VMAT techniques. The patients all had 2 cycles of carboplatin and vinorelbine before randomization
  Interventions: Drug: Navelbine; Radiation: 60 Gy/30F

INTERVENTIONS:
Drug: Navelbine — Navelbine oral 150 mg of Vinorelbine administered in 3 weekly doses a week for 6-6½ weeks
  Other Names: Vinorelbine
Radiation: 66 Gy/33F — irradiation to 66 Gy (2 Gy x 30, 5 F á weeks)
  Arms: B: 66Gy/33F+Navelbine oral 150 mg q3w
Radiation: 60 Gy/30F — irradiation to 60 Gy (2 Gy x 30, 5 F á weeks)
  Arms: A: 60Gy/30F+Navelbine oral 150 mg q3w

SUMMARY:
This study is an open label randomized multi-centre phase II trial in patients with inoperable locally advanced stage IIB-IIIB Non Small Cell Lung Cancer who fulfils the general criteria for curatively intended irradiation. The treatment plan consists of two courses of inductions chemotherapy followed of concomitant therapy chemo-radiotherapy 3 weeks after day 1 of the last induction chemotherapy has been given. The patients will be included in the study after completing the induction chemotherapy. Randomization will take place only if an acceptable dose plan can be obtained.

DETAILED DESCRIPTION:
This study was an open label randomized multi-centre phase II trial in patients with inoperable locally advanced stage IIB-IIIB Non Small Cell Lung Cancer who fulfils the general criteria for curatively intended irradiation. The treatment plan consisted of two courses of inductions chemotherapy followed of concomitant therapy chemo-radiotherapy 3 weeks after day 1 of the last induction chemotherapy has been given. The patients was included in the study after completing the induction chemotherapy. Randomization took place only if an acceptable dose plan could be obtained.

Primary endpoint: local recurrence free interval

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with histologically or cytologically documented diagnosis of locally advanced NSCLC stage IIB to IIIB without pleural effusion
* Performance status 0-1 on the ECOG scale
* Weight loss ≤10% during the last 6 months
* Adequate lung function measured as FEV1 ≥1.0
* Neutrophile count ≥1.5 x 109/L and platelet count ≥100 x 109/L
* Serum bilirubin ≤1.5 upper limit of normal (ULN)
* ALAT ≤2 x ULN
* Able to comply with study and follow-up procedures
* Patients with reproductive potential must use effective contraception
* Written (signed) informed consent to participate in the study

Exclusion Criteria:

* Any unstable systemic disease (including active infection, unstable angina, congestive heart failure, severe hepatic, renal, or metabolic disease)
* Any other active malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer)
* Prior chemotherapy for lung cancer, including neo- and adjuvant chemotherapy
* Inability to take oral medication, or requirement of intravenous alimentation
* Active peptic ulcer disease
* Nursing mothers

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olfred Hansen, MD, Principal Investigator — Odense University Hospital
Locations (6):
- Denmark (6):
  - Department of Oncology, Aalborg University Hospital, Aalborg
  - Department of Oncology, Aarhus University Hospital, Aarhus
  - Department of Oncology, Copenhagen University Hospital Herlev, Herlev
  - Department of Oncology, Odense University Hospital, Odense
  - Laboratory of Radiation Physics, Odense
  - Department of Oncology, Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: Undecided
Further studies on toxicity profiles and PET may be performed

REFERENCES:
- [Result] Hansen O, Knap MM, Khalil A, Nyhus CH, McCulloch T, Holm B, Brink C, Hoffmann L, Schytte T. A randomized phase II trial of concurrent chemoradiation with two doses of radiotherapy, 60Gy and 66Gy, concomitant with a fixed dose of oral vinorelbine in locally advanced NSCLC. Radiother Oncol. 2017 May;123(2):276-281. doi: 10.1016/j.radonc.2017.03.017. Epub 2017 Apr 11. PMID 28410809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 117 included July 2009 to August 2013
Groups:
- B: 66Gy/33F+Navelbine Oral 150 mg q3w: Navelbine oral 150 mg of Vinorelbine administered in 3 weekly doses a week for 6-6½ weeks concomitant with curatively intended irradiation to 66 Gy (2 Gy x 30, 5 F á weeks).
  Radiation technique: 3D, 4D og VMAT techniques. The patients all had 2 cycles of carboplatin and vinorelbine before randomization
  Navelbine: Navelbine oral 150 mg of Vinorelbine administered in 3 weekly doses a week for 6-6½ weeks
  66 Gy/33F: irradiation to 66 Gy (2 Gy x 30, 5 F á weeks)
Period: Overall Study
Arm/Group | B: 66Gy/33F+Navelbine Oral 150 mg q3w | A: 60Gy/30F+Navelbine Oral 150 mg q3w
Started | 58 | 59
Completed | 58 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B: 66Gy/33F+Navelbine Oral 150 mg q3w | A: 60Gy/30F+Navelbine Oral 150 mg q3w | Total
Number analyzed (Participants) | 58 | 59 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 22 | 54
  >=65 years | 26 | 37 | 63
Age, Continuous [Median (Full Range); unit: years] | 64.56 [44.38 to 79.39] | 66.63 [44.68 to 81.98] | 65.53 [44.38 to 81.98]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 36 | 62
  Male | 32 | 23 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 58 | 59 | 117

OUTCOME MEASURES:

1. Primary Outcome: Local Failure Free Survival
Description: Local failure free survival 9 month after first RT treatment measured by CT/FDG-CT
Time Frame: 9 months
Population: Analyzed as intention to treat
Measure: Median (Full Range); unit: months
Arm/Group | B: 66Gy/33F+Navelbine Oral 150 mg q3w | A: 60Gy/30F+Navelbine Oral 150 mg q3w
Number analyzed (Participants) | 58 | 59
months | 9.4 [2.8 to 67] | 9.9 [2.6 to 54]

2. Secondary Outcome: Number of Participants Who Experienced Early Toxicity to Concurrent Vinorelbine and Radiotherapy
Time Frame: 9 months
Population: Dysphagia, weight loss ≥20%, pulmonary toxicity grade 3, leucopenia grade 3 or higher
Measure: Number; unit: participants
Arm/Group | B: 66Gy/33F+Navelbine Oral 150 mg q3w | A: 60Gy/30F+Navelbine Oral 150 mg q3w
Number analyzed (Participants) | 58 | 59
participants
  Dysphagia g3+ | 7 | 6
  Pulmonary tox | 14 | 11
  Leucopenia g3+ | 4 | 3

3. Secondary Outcome: Local Tumour Control
Description: Loco-regional control
Time Frame: 9 months
Reporting Status: Not Posted, anticipated posting 2022-09

4. Secondary Outcome: Overall Survival
Description: Overall survival, death of any cause
Time Frame: 72 months
Population: Overall survival, intention to treat
Measure: Median (Full Range); unit: Months
Arm/Group | B: 66Gy/33F+Navelbine Oral 150 mg q3w | A: 60Gy/30F+Navelbine Oral 150 mg q3w
Number analyzed (Participants) | 58 | 59
Months | 25.3 [3.0 to 68] | 23.3 [3.2 to 65.6]

5. Secondary Outcome: Late Toxicity
Description: Late toxicity related to concurrent Vinorelbine and radiotherapy
Time Frame: 48 months
Reporting Status: Not Posted, anticipated posting 2022-09

6. Secondary Outcome: Disease Free Survival
Description: Disease free survival, death of any cause
Time Frame: 72 months
Measure: Median (Full Range); unit: Months
Arm/Group | B: 66Gy/33F+Navelbine Oral 150 mg q3w | A: 60Gy/30F+Navelbine Oral 150 mg q3w
Number analyzed (Participants) | 58 | 59
Months | 8.4 [.2 to 68] | 8.8 [.2 to 54]

ADVERSE EVENTS:
Time Frame: 5 years, death or recurrence
Arm/Group | B: 66Gy/33F+Navelbine Oral 150 mg q3w | A: 60Gy/30F+Navelbine Oral 150 mg q3w
All-Cause Mortality (participants affected / at risk) | 41/58 | 44/59
Serious Adverse Events (participants affected / at risk) | 18/58 | 15/59
Other Adverse Events (participants affected / at risk) | 25/58 | 20/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B: 66Gy/33F+Navelbine Oral 150 mg q3w (N=58) | A: 60Gy/30F+Navelbine Oral 150 mg q3w (N=59)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 7 (7) — Pneumonitis, pneumonia, embolus
Dysphagia (Gastrointestinal disorders) | 8 (8) | 8 (8) — Dysphagia, esophagitis, stenosis, obstipation, nausea
Herpes zoster (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Herpes zoster
Atrial fibrilation (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Atrial flutter
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B: 66Gy/33F+Navelbine Oral 150 mg q3w (N=58) | A: 60Gy/30F+Navelbine Oral 150 mg q3w (N=59)
Leucopenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 7 (7) | 6 (6)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No